CLINICAL TRIAL: NCT02964221
Title: Assessing Postoperative Cognitive Changes After Major Joint Arthroplasty: A Feasibility Study Using the CogState Brief Battery
Brief Title: Cognitive Changes After Major Joint Replacement
Acronym: Cognigram
Status: Completed | Type: Observational
Sponsor: Dr. Stephen Choi (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Choi, Assistant Professor, University of Toronto; Staff Anesthesiologist and Director of Clinical Research, Department of Anesthesia, Sunnybrook Health Sciences Centre, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 045-2015
Record Dates: First submitted 2016-11-01; First posted 2016-11-16 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Cognitive Dysfunction; Mild Cognitive Impairment; Delirium; Cognitive Deficit; Cognitive Change; Working Memory
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction; Delirium; Cognition Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cognitive Testing — Computerized CogState Brief Battery (CBB), Cognigram, assesses changes in four cognitive domains including psychomotor function, attention, learning and memory, and working memory. The CBB is a computerized test based on card games that can be administered online. .

SUMMARY:
Patients assume that cognitive performance rapidly returns to baseline after anesthesia and surgery. Several studies have shown that one week after major non-cardiac surgery about 27% of patients have postoperative cognitive dysfunction (POCD) and 10% of patients at 3 months. Very few studies have assessed the incidence of POCD beyond 3 months. POCD significantly reduces quality of life. Identifying risk factors for POCD is important because it is associated with prolonged hospital stay, loss of independence, and premature retirement. There is an urgent need to measure and document the level of cognitive change associated with surgery with an easy to use tool, both prior to admission and after discharge. This information can be used to plan appropriate care paths and to identify or test the efficacy of potential new treatments to alter the negative trajectory.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is thought to affect a significant proportion of patients after major surgery (up to 10% at 3 months). This is potentially a major public health issue because patients with POCD have prolonged hospital admission, loss of independence and mortality. Undoubtedly, if POCD is as prevalent and devastating as has been previously reported, the decision to undergo elective surgery should be influenced by the risk of developing POCD. Given the scope of the issue, the deficiencies in the literature surrounding POCD are concerning. There are many methodological issues with previous studies and the diagnosis of POCD in the perioperative period.

It is imperative that the true natures of postoperative cognitive changes are elucidated so that preoperative risk stratification can be appropriately determined. This will lead to care pathways and interventions that can modify any possible downward changes thereby reducing the negative impact on patients and the health care system.

Study Hypothesis: The incidence of postoperative cognitive changes in the joint arthroplasty population is influenced by postoperative complications, pre-existing mild cognitive impairment, and pre-existing comorbid conditions.

Study Objectives:

1. To conduct a pilot study for six to 12 months to assess both the rate of recruitment (goal of 15 participants/month) and postoperative in-person follow-up (at 6 weeks and 4.5 months), and determine if a large-scale study of 600 participants is feasible
2. To determine the sensitivity and accuracy of Cognigram (CogState Brief Battery - CBB) for detecting changes in cognitive function during the perioperative period
3. To determine whether pre-existing mild cognitive impairment (MCI), preoperative chronic inflammatory states, and acute postoperative complications affect changes in postoperative cognitive function

ELIGIBILITY:
Inclusion Criteria:

• All patients ≥ 50 years of age undergoing elective total hip or knee arthroplasty at Sunnybrook Health Sciences Centre

Exclusion Criteria:

* Lack of informed consent
* Inability to comply with study procedures or follow-up visits
* Patients with diagnosed dementia or those being treated with donepezil (Aricept®)
* Patients with severe cognitive impairment defined as baseline with a CBB score of equal to or less than 80 in at least one of the 4 CBB domains
* Patients with psychiatric diagnoses including schizophrenia, bipolar disorder, major depressive mood disorder
* Patients undergoing a second joint replacement & previously enrolled in this study within the past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthroplasty (THA) or total knee arthroplasty (TKA) at the Holland Orthopedic and Arthritic Centre (HOAC) at Sunnybrook Health Sciences Centre (SHSC).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Brief Battery (CBB) score from baseline to 4.5 months after surgery | 4.5 months after surgery
  Change in Cognitive Brief Battery (CBB) score from baseline to 4.5 months after surgery

SECONDARY OUTCOMES:
Proportion of patients developing severe cognitive dysfunction at 4.5 months after surgery (defined as CBB score less than 80) | 4.5 months after surgery
  Proportion of patients developing severe cognitive dysfunction at 4.5 months after surgery (defined as CBB score less than 80)
Proportion of patients developing mild cognitive impairment at 4.5 months after surgery defined as CBB score between 81 and 90 | 4.5 months after surgery
  Proportion of patients developing mild cognitive impairment at 4.5 months after surgery defined as CBB score between 81 and 90
The effect of pre-operative mild cognitive impairment, pre-operative chronic inflammatory states, postoperative delirium, and postoperative complications on the incidence of mild cognitive impairment and severe cognitive dysfunction at 4.5 months | 4.5 months after surgery
  The effect of pre-operative mild cognitive impairment, pre-operative chronic inflammatory states, postoperative delirium, and postoperative complications on the incidence of mild cognitive impairment and severe cognitive dysfunction at 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD,FRCPC,MSc, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: Undecided